CLINICAL TRIAL: NCT05493982
Title: Evaluation of the Be Vape Free Curriculum of the Tobacco Prevention Toolkit
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bonnie Halpern-Felsher, Marron and Mary Elizabeth Kendrick Professor in Pediatrics II, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 61965; 1R01CA263121 (NIH)
Record Dates: First submitted 2022-08-06; First posted 2022-08-09 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-07

CONDITIONS: E-cigarette Use
Keywords: youth; tobacco; education; health; prevention; vaping; e-cigarette
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Receives Stanford vaping prevention curriculum (pilot phase) (Experimental): Stanford vaping prevention curriculum is administered as pilot arm preceding main experimental intervention.
  Interventions: Behavioral: Stanford Vaping Prevention curriculum
- Receives Stanford vaping prevention curriculum (randomized phase) (Experimental): Stanford vaping prevention curriculum is administered.
  Interventions: Behavioral: Stanford Vaping Prevention curriculum
- Does not receive Stanford vaping prevention curriculum (randomized phase) (No Intervention): Receives another curriculum or no vaping prevention education.

INTERVENTIONS:
Behavioral: Stanford Vaping Prevention curriculum — Stanford vaping prevention curriculum delivered as a 5-session course administered in a school classroom setting.
  Arms: Receives Stanford vaping prevention curriculum (pilot phase); Receives Stanford vaping prevention curriculum (randomized phase)

SUMMARY:
The Stanford Tobacco Prevention Toolkit is a free online curriculum developed for use by educators and health professionals in providing tobacco-specific prevention education to middle and high school students. A set of lessons focused on e-cigarette/vaping prevention education specifically is called the Be Vape Free curriculum. The aims of this study are to determine: (1) whether the Be Vape Free curriculum is effective in increasing middle and high school students' resistance to using tobacco and in decreasing positive attitudes towards and intentions to use e-cigarettes; (2) whether the Curriculum is effective in changing middle and high school students' actual use of tobacco; and (3) Examine heterogenous treatment effects identifying groups that benefit the most and those who do not benefit at all from the intervention.

ELIGIBILITY:
Inclusion Criteria:

Middle school and high school students receiving health education at schools participating in the study

Exclusion Criteria:

None

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10800 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in e-cigarette use | Change from baseline to follow-up at approximately 156 weeks
  Investigator-originated survey measures (questions) assess ever e-cigarette use & past 30-day tobacco use. This outcome measure assesses e-cigarette use.
Change in intention to use of e-cigarettes scaled score as measured by investigator-originated survey | Change from baseline to follow-up at approximately 156 weeks
  This survey measures change in intention to use e-cigarettes with questions related to the participant's knowledge of and resistance to use of e-cigarettes.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Halpern-Felsher, Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No